CLINICAL TRIAL: NCT02421224
Title: Social and Monetary Incentives for Smoking Cessation at Large Employers
Acronym: SMILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH); Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UCaliforniaBerkeley; 5R01DA035384 (NIH)
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Tobacco Use Disorder
Keywords: Smoking Cessation; Incentives; Health Behavior; Smoking; Work-site
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Health Behavior; Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- Usual Care (Active Comparator): Participants will receive in-person group counseling from a trained smoking cessation counselor. Participants will learn about reasons to quit smoking, strategies for quitting smoking, and additional resources available to support the quit attempt. Participants will also complete a quit plan.
  Interventions: Behavioral: Usual Care
- Deposits (Experimental): Same as Usual Care, plus participants will have to deposit a certain amount of their own money as an incentive to quit smoking. Participants will be able to make additional voluntary deposits above the minimum amount. The participant will be refunded all deposits if he quits smoking at 3 months, as verified by a urine cotinine test. The participant will forfeit all deposits if he continues to smoke at 3 months, as verified by a urine cotinine test.
  Interventions: Behavioral: Usual Care; Behavioral: Deposits
- Small Individual Bonus (Experimental): Same as Usual Care, plus each participant will receive a monetary bonus from the study investigators if he or she quit smoking, as verified by a urine cotinine test.
  Interventions: Behavioral: Usual Care; Behavioral: Small Individual Bonus
- Large Individual Bonus (Experimental): Same as Usual Care, plus each participant will receive a monetary bonus from the study investigators if he or she quit smoking, as verified by a urine cotinine test. The bonus is twice the value of that in the Small Individual Bonus group.
  Interventions: Behavioral: Usual Care; Behavioral: Large Individual Bonus
- Team Bonus (Experimental): Same as Usual Care, plus each participant will be randomly assigned one teammate to provide social support during the quit attempt. If the participant and assigned teammate both quit smoking at 3 months, as verified by a urine cotinine test, then each will receive a monetary bonus. The team bonus is equal in value to that in the Large Individual Bonus group.
  Interventions: Behavioral: Usual Care; Behavioral: Teammate; Behavioral: Team Bonus
- Deposits plus Small Individual Bonus (Experimental): Same as Usual Care, plus the participant will follow the protocol for deposits as described for the Deposits group and will follow the protocol for the monetary bonus as described for the Small Individual Bonus group.
  Interventions: Behavioral: Usual Care; Behavioral: Deposits; Behavioral: Small Individual Bonus
- Deposits plus Large Individual Bonus (Experimental): Same as Usual Care, plus the participant will follow the protocol for deposits as described for the Deposits group and will follow the protocol for the monetary bonus as described for the Large Individual Bonus group.
  Interventions: Behavioral: Usual Care; Behavioral: Deposits; Behavioral: Large Individual Bonus
- Deposits plus Teammate (Experimental): Same as Usual Care, plus the participant will follow the protocol for deposits as described for the Deposits group and will be randomly assigned one other participant to serve as a teammate who provides social support during the quit attempt.
  Interventions: Behavioral: Usual Care; Behavioral: Deposits; Behavioral: Teammate
- Deposits plus Team Bonus (Experimental): Same as Usual Care, plus the participant will follow the protocol for deposits as described for the Deposits group, will be randomly assigned a teammate, and will follow the protocol for the monetary bonus as described for the Team Bonus group.
  Interventions: Behavioral: Usual Care; Behavioral: Deposits; Behavioral: Teammate; Behavioral: Team Bonus

INTERVENTIONS:
Behavioral: Usual Care — Participants will receive in-person group counseling from a trained smoking cessation counselor. Participants will learn about reasons to quit smoking, strategies for quitting smoking, and additional resources available to support the quit attempt. Participants will also complete a quit plan.
Behavioral: Deposits — Participants will have to deposit a certain amount of their own money at enrollment. Participants will be able to make additional voluntary deposits above the minimum amount during the intervention period. The participant will be refunded all deposits if he quits smoking at 3 months, as verified by a urine cotinine test. The participant will forfeit all deposits if he continues to smoke at 3 months, as verified by a urine cotinine test.
  Arms: Deposits; Deposits plus Large Individual Bonus; Deposits plus Small Individual Bonus; Deposits plus Team Bonus; Deposits plus Teammate
Behavioral: Small Individual Bonus — Each participant will receive a monetary bonus from the study investigators if he or she quit smoking, as verified by a urine cotinine test.
  Arms: Deposits plus Small Individual Bonus; Small Individual Bonus
Behavioral: Large Individual Bonus — Each participant will receive a monetary bonus from the study investigators if he or she quit smoking, as verified by a urine cotinine test. The bonus is twice the value of that in the Small Individual Bonus group.
  Arms: Deposits plus Large Individual Bonus; Large Individual Bonus
Behavioral: Teammate — Each participant will be randomly assigned one teammate to provide social support during the quit attempt. Each participant will be assigned to a participating coworker who speaks the same primary language and works the same work shift as the participant.
  Arms: Deposits plus Team Bonus; Deposits plus Teammate; Team Bonus
Behavioral: Team Bonus — If the participant and assigned teammate both quit smoking at 3 months, as verified by a urine cotinine test, then each will receive a monetary bonus. The team bonus is equal in value to that in the Large Individual Bonus group.
  Arms: Deposits plus Team Bonus; Team Bonus

SUMMARY:
The investigators will conduct a cluster randomized controlled trial of several behavioral interventions for smoking cessation among a sample of employees at large workplaces in the Bangkok metropolitan area. The study aims to test the impacts of different incentive structures for smoking cessation on take-up, effectiveness, and cost-effectiveness. The interventions are designed to elucidate certain principles from the field of behavioral economics.

ELIGIBILITY:
Inclusion Criteria:

* Current full-time employee of a participating company
* Smoker of 100+ cigarettes during lifetime
* Smoker of 10+ cigarettes per week
* Individual is aged 18+ years old
* Smoker wants to quit within the next 6 months

Exclusion Criteria:

* Expects to leave company within the next 12 months
* Is currently pregnant
* Are unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4190 (Actual)
Dates: Start 2015-04; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William H. Dow, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- Mahidol University, Bangkok, Thailand

REFERENCES:
- [Result] White JS, Lowenstein C, Srivirojana N, Jampaklay A, Dow WH. Incentive programmes for smoking cessation: cluster randomized trial in workplaces in Thailand. BMJ. 2020 Oct 14;371:m3797. doi: 10.1136/bmj.m3797. PMID 33055176

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Worksites
Groups:
- Deposits Plus Team Bonus: Same as Usual Care, plus the participant will follow the protocol for deposits as described for the Deposits group, will be randomly assigned a teammate, and will follow the protocol for the monetary bonus as described for the Team Bonus group.
  Usual Care: Participants will receive in-person group counseling from a trained smoking cessation counselor. Participants will learn about reasons to quit smoking, strategies for quitting smoking, and additional resources available to support the quit attempt. Participants will also complete a quit plan.
  Deposits: Participants will have to deposit a certain amount of their own money at enrollment. Participants will be able to make additional voluntary deposits above the minimum amount during the intervention period. The participant will be refunded all deposits if he quits smoking at 3 months, as verified by a urine test. The participant will forfeit all deposits if he continues to smoke at 3 months, as verified by a urine test.
  Teammate: Each participant will be randomly assigned one teammate to provide social support during the quit attempt. Each participant will be assigned to a participating coworker who speaks the same primary language and works the same work shift as the participant.
  Team Bonus: If the participant and assigned teammate both quit smoking at 3 mos., as verified by a urine cotinine test, then each will receive a monetary bonus. The team bonus is equal in value to that in the Large Individual Bonus group.
Period: Overall Study
Arm/Group | Usual Care | Deposits | Small Individual Bonus | Large Individual Bonus | Team Bonus | Deposits Plus Small Individual Bonus | Deposits Plus Large Individual Bonus | Deposits Plus Teammate | Deposits Plus Team Bonus
Started | 444; 12 Worksites | 397; 11 Worksites | 508; 11 Worksites | 482; 11 Worksites | 495; 11 Worksites | 515; 11 Worksites | 489; 11 Worksites | 364; 11 Worksites | 496; 12 Worksites
Completed | 442; 12 Worksites | 394; 11 Worksites | 507; 11 Worksites | 479; 11 Worksites | 491; 11 Worksites | 513; 11 Worksites | 489; 11 Worksites | 362; 11 Worksites | 495; 12 Worksites
Not Completed | 2; 0 Worksites | 3; 0 Worksites | 1; 0 Worksites | 3; 0 Worksites | 4; 0 Worksites | 2; 0 Worksites | 0; 0 Worksites | 2; 0 Worksites | 1; 0 Worksites

BASELINE CHARACTERISTICS:
Groups:
- Deposits Plus Team Bonus: Same as Usual Care, plus the participant will follow the protocol for deposits as described for the Deposits group, will be randomly assigned a teammate, and will follow the protocol for the monetary bonus as described for the Team Bonus group.
  Usual Care: Participants will receive in-person group counseling from a trained smoking cessation counselor. Participants will learn about reasons to quit smoking, strategies for quitting smoking, and additional resources available to support the quit attempt. Participants will also complete a quit plan.
  Deposits: Participants will have to deposit a certain amount of their own money at enrollment. Participants will be able to make additional voluntary deposits above the minimum amount during the intervention period. The participant will be refunded all deposits if he quits smoking at 3 months, as verified by a urine test. The participant will forfeit all deposits if he continues to smoke at 3 months, as verified by a urine test.
  Teammate: Each participant will be randomly assigned one teammate to provide social support during the quit attempt. Each participant will be assigned to a participating coworker who speaks the same primary language and works the same work shift as the participant.
  Team Bonus: If the participant and assigned teammate both quit smoking at 3 months, as verified by a urine test, then each will receive a monetary bonus. The team bonus is equal in value to that in the Large Individual Bonus group.
- Total: Total of all reporting groups
Arm/Group | Usual Care | Deposits | Small Individual Bonus | Large Individual Bonus | Team Bonus | Deposits Plus Small Individual Bonus | Deposits Plus Large Individual Bonus | Deposits Plus Teammate | Deposits Plus Team Bonus | Total
Number analyzed (Participants) | 444 | 397 | 508 | 482 | 495 | 515 | 489 | 364 | 496 | 4190
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Number analyzed includes those in the primary analysis, dropping those who died before the primary endpoint and those who were missing at least one covariate in the regression analyses.
  years
    number analyzed (Participants) | 442 | 394 | 507 | 479 | 491 | 513 | 489 | 362 | 495 | 4172
    (all) | 32 [26 to 39] | 32 [27 to 40] | 31 [26 to 38] | 33 [27 to 42] | 30 [25 to 38] | 34 [27 to 40] | 31 [25 to 38] | 35 [28 to 42] | 32 [25 to 40] | 32 [26 to 40]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number analyzed includes those in the primary analysis, dropping those who died before the primary endpoint and those who were missing at least one covariate in the regression analyses.
  Participants
    number analyzed (Participants) | 442 | 394 | 507 | 479 | 491 | 513 | 489 | 362 | 495 | 4172
    Female | 3 | 18 | 20 | 4 | 2 | 10 | 25 | 15 | 9 | 106
    Male | 439 | 376 | 487 | 475 | 489 | 503 | 464 | 347 | 486 | 4066
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Thailand | 444 | 397 | 508 | 482 | 495 | 515 | 489 | 364 | 496 | 4190

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Smoking Abstinence at 12 Months
Description: 7-day point prevalence of abstinence measured 12 months after enrollment using self-reported abstinence and urine cotinine test results
Time Frame: 12 months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Deposits | Small Individual Bonus | Large Individual Bonus | Team Bonus | Deposits Plus Small Individual Bonus | Deposits Plus Large Individual Bonus | Deposits Plus Teammate | Deposits Plus Team Bonus
Number analyzed (Participants) | 442 | 394 | 507 | 479 | 491 | 513 | 489 | 362 | 495
Participants | 42 | 57 | 74 | 104 | 60 | 72 | 91 | 49 | 67

2. Secondary Outcome: Proportion of Participants With Smoking Abstinence at 3 Months
Description: 7-day point prevalence of abstinence measured 3 months after enrollment based on self-reported abstinence and urine cotinine test results
Time Frame: 3 months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Deposits | Small Individual Bonus | Large Individual Bonus | Team Bonus | Deposits Plus Small Individual Bonus | Deposits Plus Large Individual Bonus | Deposits Plus Teammate | Deposits Plus Team Bonus
Number analyzed (Participants) | 442 | 394 | 507 | 479 | 491 | 513 | 489 | 362 | 495
Participants | 40 | 61 | 64 | 88 | 56 | 66 | 89 | 38 | 73

3. Secondary Outcome: Program Acceptance
Description: Proportion of eligible smokers who consent to participate in the main intervention
Time Frame: At 0 months (at enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Deposits | Small Individual Bonus | Large Individual Bonus | Team Bonus | Deposits Plus Small Individual Bonus | Deposits Plus Large Individual Bonus | Deposits Plus Teammate | Deposits Plus Team Bonus
Number analyzed (Participants) | 442 | 394 | 507 | 479 | 491 | 513 | 489 | 362 | 495
Participants | 271 | 202 | 345 | 290 | 293 | 270 | 279 | 173 | 328

4. Secondary Outcome: Proportion of Participants With Smoking Abstinence at 6 Months
Description: 7-day point prevalence of abstinence measured 6 months after enrollment based on self-reported abstinence and urine cotinine test results
Time Frame: 6 months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Deposits | Small Individual Bonus | Large Individual Bonus | Team Bonus | Deposits Plus Small Individual Bonus | Deposits Plus Large Individual Bonus | Deposits Plus Teammate | Deposits Plus Team Bonus
Number analyzed (Participants) | 442 | 394 | 507 | 479 | 491 | 513 | 489 | 362 | 495
Participants | 48 | 54 | 62 | 104 | 52 | 67 | 106 | 48 | 72

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Deposits: Same as Usual Care, plus participants will have to deposit a certain amount of their own money as an incentive to quit smoking. Participants will be able to make additional voluntary deposits above the minimum amount. The participant will be refunded all deposits if he quits smoking at 3 months, as verified by a urine cotinine test. The participant will forfeit all deposits if he continues to smoke at 3 months, as verified by a urine cotinine test.
  Usual Care: Same as Usual Care only group.
  Deposits: Participants will have to deposit a certain amount of their own money at enrollment. Participants will be able to make additional voluntary deposits above the minimum amount during the intervention period. The participant will be refunded all deposits if he quits smoking at 3 months, as verified by a urine cotinine test. The participant will forfeit all deposits if he continues to smoke at 3 months, as verified by a urine cotinine test.
- Small Individual Bonus: Same as Usual Care, plus each participant will receive a monetary bonus from the study investigators if he or she quit smoking, as verified by a urine cotinine test.
  Usual Care: Same as Usual Care only group.
  Small Individual Bonus: Each participant will receive a monetary bonus from the study investigators if he or she quit smoking, as verified by a urine cotinine test.
- Large Individual Bonus: Same as Usual Care, plus each participant will receive a monetary bonus from the study investigators if he or she quit smoking, as verified by a urine cotinine test. The bonus is twice the value of that in the Small Individual Bonus group.
  Usual Care: Same as Usual Care only group.
  Large Individual Bonus: Each participant will receive a monetary bonus from the study investigators if he or she quit smoking, as verified by a urine cotinine test. The bonus is twice the value of that in the Small Individual Bonus group.
- Team Bonus: Same as Usual Care, plus each participant will be randomly assigned one teammate to provide social support during the quit attempt. If the participant and assigned teammate both quit smoking at 3 months, as verified by a urine cotinine test, then each will receive a monetary bonus. The team bonus is equal in value to that in the Large Individual Bonus group.
  Usual Care: Same as Usual Care only group.
  Teammate: Each participant will be randomly assigned one teammate to provide social support during the quit attempt. Each participant will be assigned to a participating coworker who speaks the same primary language and works the same work shift as the participant.
  Team Bonus: If the participant and assigned teammate both quit smoking at 3 months, as verified by a urine cotinine test, then each will receive a monetary bonus. The team bonus is equal in value to that in the Large Individual Bonus group.
- Deposits Plus Small Individual Bonus: Same as Usual Care, plus the participant will follow the protocol for deposits as described for the Deposits group and will follow the protocol for the monetary bonus as described for the Small Individual Bonus group.
  Usual Care: Same as Usual Care only group.
  Deposits: Participants will have to deposit a certain amount of their own money at enrollment. Participants will be able to make additional voluntary deposits above the minimum amount during the intervention period. The participant will be refunded all deposits if he quits smoking at 3 months, as verified by a urine cotinine test. The participant will forfeit all deposits if he continues to smoke at 3 months, as verified by a urine cotinine test.
  Small Individual Bonus: Each participant will receive a monetary bonus from the study investigators if he or she quit smoking, as verified by a urine cotinine test.
- Deposits Plus Large Individual Bonus: Same as Usual Care, plus the participant will follow the protocol for deposits as described for the Deposits group and will follow the protocol for the monetary bonus as described for the Large Individual Bonus group.
  Usual Care: Same as Usual Care only group.
  Deposits: Participants will have to deposit a certain amount of their own money at enrollment. Participants will be able to make additional voluntary deposits above the minimum amount during the intervention period. The participant will be refunded all deposits if he quits smoking at 3 months, as verified by a urine cotinine test. The participant will forfeit all deposits if he continues to smoke at 3 months, as verified by a urine cotinine test.
  Large Individual Bonus: Each participant will receive a monetary bonus from the study investigators if he or she quit smoking, as verified by a urine cotinine test. The bonus is twice the value of that in the Small Individual Bonus group.
- Deposits Plus Teammate: Same as Usual Care, plus the participant will follow the protocol for deposits as described for the Deposits group and will be randomly assigned one other participant to serve as a teammate who provides social support during the quit attempt.
  Usual Care: Same as Usual Care only group.
  Deposits: Same as Deposits only group.
  Teammate: Each participant will be randomly assigned one teammate to provide social support during the quit attempt. Each participant will be assigned to a participating coworker who speaks the same primary language and works the same work shift as the participant.
- Deposits Plus Team Bonus: Same as Usual Care, plus the participant will follow the protocol for deposits as described for the Deposits group, will be randomly assigned a teammate, and will follow the protocol for the monetary bonus as described for the Team Bonus group.
  Usual Care: Same as Usual Care only group.
  Deposits: Same as Deposits only group.
  Teammate: Each participant will be randomly assigned one teammate to provide social support during the quit attempt. Each participant will be assigned to a participating coworker who speaks the same primary language and works the same work shift as the participant.
  Team Bonus: If the participant and assigned teammate both quit smoking at 3 months, as verified by a urine cotinine test, then each will receive a monetary bonus. The team bonus is equal in value to that in the Large Individual Bonus group.
Arm/Group | Usual Care | Deposits | Small Individual Bonus | Large Individual Bonus | Team Bonus | Deposits Plus Small Individual Bonus | Deposits Plus Large Individual Bonus | Deposits Plus Teammate | Deposits Plus Team Bonus
All-Cause Mortality (participants affected / at risk) | 2/444 | 2/397 | 1/508 | 2/482 | 0/495 | 1/515 | 0/489 | 1/364 | 1/496
Serious Adverse Events (participants affected / at risk) | 0/444 | 0/397 | 0/508 | 0/482 | 0/495 | 0/515 | 0/489 | 0/364 | 0/496
Other Adverse Events (participants affected / at risk) | 0/444 | 0/397 | 0/508 | 0/482 | 0/495 | 0/515 | 0/489 | 0/364 | 0/496

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/24/NCT02421224/Prot_SAP_000.pdf